CLINICAL TRIAL: NCT00196417
Title: Randomized-Double Blind Trial to Assess the Incidence and Clinical Relevance of Heparin-Induced Thrombocytopenia (HIT) Antibodies in Trauma Patients Treated With Unfractionated or Low-Molecular Weight Heparin, the HIT-TRAP Trial
Brief Title: The HIT-TRAP Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Medicine Greifswald (Other)
Collaborators: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-09

CONDITIONS: Heparin-Induced Thrombocytopenia
Keywords: heparin-induced thrombocytopenia; HIT; unfractionated heparin; UFH; low-molecular-weight heparin; LMWH; thrombosis prophylaxis; HIT-antibody
MeSH Terms: interventions — Heparin, Low-Molecular-Weight

INTERVENTIONS:
Drug: Standard heparin (UFH) versus certoparin (LMWH)

SUMMARY:
Randomised, double blind trial in non-intensive care trauma patients comparing unfractionated heparin (UFH) or low-molecular-weight heparin (LMWH) in heparin-induced thrombocytopenia (HIT).

DETAILED DESCRIPTION:
This is a randomised, double blind trial including trauma patients with need for thrombosis prophylaxis with heparin. Patients receive either unfractionated heparin (UFH) or low-molecular-weight heparin (LMWH).

Heparin-induced thrombocytopenia (HIT) antibodies are measured on days 1 and 10. There are daily platelet counts. On discharge an ultrasound doppler of the lower extremities is performed to rule out deep vein thrombosis (DVT).

Three months after discharge every patient is answering a questionnaire about thromboembolic complications following discharge.

The key questions of the study are whether the two heparins cause HIT-antibodies in differing frequencies, and if yes, whether these differences lead to different clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* trauma-surgical patient
* consent given
* minimum age 18
* expected inpatient period at least 7 days
* need for thrombosis prophylaxis with heparin

Exclusion Criteria:

* intolerance of one of the study drugs
* malignancy with life expectancy < 3 months
* pregnancy/lactation
* drug or alcohol abuse
* fibrinolytic therapy
* need for extracorporal circulation (e.g. cardiopulm. bypass, hemodialysis) at study entry
* participation in another clinical trial within 30 days prior to intended inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2003-01; Study Completion 2005-11

PRIMARY OUTCOMES:
Frequency of formation of HIT-antibodies during prophylactic treatment with UFH or LMWH in trauma-surgical patients

SECONDARY OUTCOMES:
Thromboembolic complications (TECs) during inpatient period in relation to heparin received and HIT-antibody status
TECs during 3 months following discharge in relation to heparin received and HIT-antibody status

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Greinacher, Prof. Dr., Principal Investigator — Ernst-Moritz-Arndt University Greifswald, Germany
Locations (1):
- Ernst-Moritz-Arndt University, Depts. of Transfusion Medicine / Trauma surgery, Greifswald, Germany